CLINICAL TRIAL: NCT06069687
Title: A Phase 1 Open-label Intrathecal Administration of MELPIDA to Determine the Safety and Efficacy for Patients With Spastic Paraplegia Type 50 (SPG50) Caused by a Mutation in the AP4M1 Gene
Brief Title: Administration of MELPIDA to Determine the Safety and Efficacy for Patients With Spastic Paraplegia Type 50
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Gregory Costain, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000079110
Record Dates: First submitted 2023-08-17; First posted 2023-10-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Spastic Paraplegia Type 50

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MELPIDA (Experimental): A single intrathecal infusion of 10 mL at 1E14 vg/mL for a total dose of 1E15 vg (open-label)
  Interventions: Biological: MELPIDA

INTERVENTIONS:
Biological: MELPIDA — A single intrathecal infusion of 10 mL at 1E14 vg/mL for a total dose of 1E15 vg

SUMMARY:
This will be a first-in-human Phase I, open-label, single dose clinical study of MELPIDA administered intrathecally (IT) through a lumbar puncture (LP) to a single subject with confirmed pathogenic mutations in the Adaptor Related Protein Complex 4 Subunit Mu 1 (AP4M1) gene. The primary outcome will be the determination of the safety and tolerability of MELPIDA in patients with SPG50, based on development of toxicity.

The secondary outcome will be a preliminary exploration of efficacy of the treatment.

MELPIDA, is a recombinant serotype 9 adeno-associated virus (AAV) encoding a codon-optimized human AP4M1 transgene and will be administer to the patient via a single intrathecal infusion of 10 mL at 1E14 vg/mL for a total dose of 1E15 vg.

The total study duration is 5 years post dosing and the participant will be tested at screening/baseline (-28 to -7 days), return for dosing, and then follow-up visits post-dosing on Days 7 (+/-2), 30 (+/-2), 60 (+/-2), 90 (+/-14), 180 (+/-14), 270 (+/-14), 360 (+/-14), 540 (+/-14), and 720 (+/-14) days, then annually for the last 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age < 5 years old
* Confirmed diagnosis of SPG50 disease by:
* Genomic DNA mutation analysis demonstrating homozygous or compound heterozygous, pathogenic and/or potentially pathogenic variants in the AP4M1 gene
* Clinical history or examination features consistent with SPG50 and that include neurologic dysfunction
* Parent/legal guardian willing to provide written informed consent for their child prior to participation in the study
* Subject able to comply with all protocol requirements and procedures

Exclusion Criteria:

* Inability to participate in study procedures (as determined by the site investigator)
* Presence of a concomitant medical condition that precludes lumbar puncture (LP) or use of anesthetics
* History of bleeding disorder or any other medical condition or circumstance in which lumbar puncture is contraindicated according to local institutional policy
* Inability to be safely sedated in the opinion of the clinical anesthesiologist
* Active infection, at the time of dosing, based on clinical observations
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer
* Inability of the patient to undergo MRI according to local institutional policy
* Inability of the patient to undergo any other procedure required in this study
* The presence of significant non-SPG50 related central nervous system (CNS) impairment or behavioral disturbances that would confound the scientific rigor or interpretation of results of the study
* Have received an investigational drug within 30 days prior to screening or plan to receive an investigational drug (other than gene therapy) during the study.
* Enrollment and participation in another interventional clinical trial
* Contraindication to MELPIDA or any of its ingredients
* Contraindication to any of the immune suppression medications used in this study
* Clinically significant abnormal laboratory values (GGT, ALT, and AST, or total bilirubin > 3 × Upper Limit of Normal (ULN), creatinine ≥ 1.5 mg/dL, hemoglobin [Hgb] < 6 or > 20 g/dL; white blood cell (WBC) > 20,000 per cmm) prior to gene replacement therapy. Patients with an elevated bilirubin level that is unequivocally the result of neonatal jaundice shall not be excluded

Ages: 0 Years to 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of unanticipated anticipated treatment-related toxicities, Grade 3 or higher | through study completion, an average of 5 years
  collection of occurrence and severity of serious adverse events. Incidence of serious adverse events and adverse events throughout the study, as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Higher grade values indicated greater severity. Grade 1 - Grade 5.
Change from baseline in nerve conduction velocity | Screening, Day 21, and Month 3, 6, 12, 24, 36, 48 and 60
  Nerve conduction studies will be used to determine nerve conduction velocity. Nerve conduction studies involve providing a small electrical stimulus to either a motor or sensor nerve and then measuring the resulting action potential at distal point of that nerve (for sensory nerve studies) or at the muscle that the nerve innervates (motor nerve studies). Velocity of conduction (measured between the two points and represented in m/s) will be obtained. The value is compared to standard reference values for age.
Determination of liver safety | Screening, Month 6, 12, 24, 36, 48 and 60
  Changes in Liver Ultrasound findings from baseline. Incidence of serious adverse events and adverse events throughout the study, as assessed by CTCAE v5.0
Determination of liver safety | Screening, Day -1, 2, 7, 14, 21 and 28, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60
  Liver laboratory test: alanine transaminase (ALT) in U/L
Determination of liver safety | Screening, Day -1, 2, 7, 14, 21 and 28, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60
  Liver laboratory test: aspartate aminotransferase (AST) in U/L
determination of liver safety | Screening, Day -1, 2, 7, 14, 21 and 28, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60
  Liver laboratory test: Total bilirubins in umol/L
Determination of liver safety | Screening, Day -1, 2, 7, 14, 21 and 28, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60
  Liver laboratory test: direct bilirubins in umol/L
Determination of liver safety | Screening, Day -1, 2, 7, 14, 21 and 28, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60
  Liver laboratory test: alkaline phosphatase (ALP) in U/L
Determination of liver safety | Screening, Day -1, 2, 7, 14, 21 and 28, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60
  Liver laboratory test: gamma-glutamyl transferase (GGT) in U/L
Change from baseline in nerve conduction amplitude | Screening, Day 21, and Month 3, 6, 12, 24, 36, 48 and 60
  Nerve conduction study will be done to assess nerve conduction amplitude. Nerve conduction studies involve providing a small electrical stimulus to either a motor or sensor nerve and then measuring the resulting action potential at distal point of that nerve (for sensory nerve studies) or at the muscle that the nerve innervates (motor nerve studies). Amplitude of the action potential (measured at the distal site and represented in uV for sensory amplitudes and mV for motor amplitudes) will be obtained. The value is compared to standard reference values for age.

SECONDARY OUTCOMES:
Stability or improvement in spasticity | Screening, Day -1, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60.
  Modified Ashworth scale (0-4). 0: no increase in muscle tone; 1: slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension; 1+: slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of motion; 2: more marked increase in muscle tone through most of the range of motion, but affected part(s) easily moved; 3: considerable increase in muscle tone, passive movement difficult; 4: affected part(s) rigid in flexion or extension. Values reported separately for right and left upper and lower limbs.
Stability or improvement in spasticity | Screening, Day -1, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60.
  Tardieu scale (0-5). 0: no resistance throughout passive movement; 1: slight resistance throughout with no clear catch at a precise angle; 2: clear catch at a precise angle, followed by release; 3: fatiguable clonus (<10 seconds) occurring at a precise angle; 4: unfatiguable clonus (>10 seconds) occurring at a precise angle; 5: joint immobile. Values reported separately for right and left upper and lower limbs.

OTHER OUTCOMES:
Motor function, neuropsychological, and disease burden assessments | Screening, Day -1, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60.
  Bayley 4 (Fine Motor, Gross Motor, Cognitive & Language). Scores are aggregated for each domain into a scaled score. The highest possible score on a subtest or subdomain is 19, and the lowest possible score is 1. Scores from 8 to 12 are considered average.
Motor function, neuropsychological, and disease burden assessments | Screening, Day -1, 7, 14, 21 and 28, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60.
  Number of seizures per day (numerical value)
Motor function, neuropsychological, and disease burden assessments | Screening, Day -1, 7, 14, 21 and 28, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60.
  Type of seizures, if applicable
Motor function, neuropsychological, and disease burden assessments | Screening, Day -1, 7, 14, 21 and 28, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60.
  Seizure triggers, if applicable.
  Trigger will be defined by any observer or the participant. An open answer format will be collected.
Motor function, neuropsychological, and disease burden assessments | Screening, Day -1, 7, 14, 21 and 28, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60.
  Seizure rescue medication used, if applicable
Motor function, neuropsychological, and disease burden assessments | Screening, Day -1, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60.
  Clinical Global Impression of Overall Change by Physician (1-7); 1: very much improved to 7: very much worse. Single value reported.
Motor function, neuropsychological, and disease burden assessments | Screening, Day -1, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60.
  Vineland (Comprehensive Parent/Caregiver Form). The domain scores are expressed as standard scores with a mean of 100 and standard deviation of 15; domains: communication, daily living skills, socialization and motor skills.
motor function, neuropsychological, and disease burden assessments | Screening, Day -1, 7, 14, 21 and 28, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60.
  Number of falls per day
Motor function, neuropsychological, and disease burden assessments | Screening, Day -1, 7, 14, 21 and 28, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60.
  Causes of any falls reported, as applicable
Motor function, neuropsychological, and disease burden assessments | Screening, Day -1, and Month 3, 6, 9, 12, 18, 24, 36, 48 and 60.
  Clinical Severity of Illness by Physician (1-7); 1: normal, shows no sign of illness to 7: among the most extremely ill of patients. Single value reported.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dowling JJ, Pirovolakis T, Devakandan K, Stosic A, Pidsadny M, Nigro E, Sahin M, Ebrahimi-Fakhari D, Messahel S, Varadarajan G, Greenberg BM, Chen X, Minassian BA, Cohn R, Bonnemann CG, Gray SJ. AAV gene therapy for hereditary spastic paraplegia type 50: a phase 1 trial in a single patient. Nat Med. 2024 Jul;30(7):1882-1887. doi: 10.1038/s41591-024-03078-4. Epub 2024 Jun 28. PMID 38942994